CLINICAL TRIAL: NCT01605253
Title: Eszopiclone for the Treatment of PTSD
Brief Title: Eszopiclone for the Treatment of Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R34MH091338-01A1 (NIH); 1R34MH091338-01A1 (NIH)
Record Dates: First submitted 2012-05-10; First posted 2012-05-24 (Estimated); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-11

CONDITIONS: Posttraumatic Stress Disorders
Keywords: Post-traumatic stress disorder; sleep disturbance; insomnia; cytokines; anxiety; traumatic event; memory
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Parasomnias; Sleep Initiation and Maintenance Disorders; Anxiety Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eszopiclone (Active Comparator): The total study duration is 16 weeks, with subjects taking 3mg eszopiclone at bedtime for 12 weeks. There is one follow-up visit after the 12 week treatment phase.
  Interventions: Drug: Eszopiclone
- Placebo (Placebo Comparator): The total study duration is 16 weeks, with subjects taking placebo at bedtime for 12 weeks. There is one follow-up visit after the 12 week treatment phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — Eszopiclone has been approved by the US Food and Drug Administration (FDA) for the treatment of insomnia (inability to sleep). Eszopiclone has not been specifically approved by the FDA for people who have PTSD-related sleep disturbance.
  Other Names: Lunesta®
  Arms: Eszopiclone
Drug: Placebo — The placebo used in this study looks exactly like eszopiclone but contains no active ingredients.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if eszopiclone relative to placebo (sugar pill) is effective and tolerable for people with posttraumatic stress disorder (PTSD)-related sleep disturbance. The investigators will also examine the impact of treatment on sleep patterns, memory recall bias, and level of inflammatory markers (cytokines). The investigators predict eszopiclone will lead to greater improvement than placebo in measures of PTSD symptoms, memory recall bias, and level of inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients age 18-65 with a primary diagnosis of PTSD and associated sleep disturbance
* Good physical health
* Willingness and ability to comply with the requirements of the study protocol

Exclusion Criteria:

* Women pregnant, lactating, or of childbearing potential not using medically accepted contraception
* Concurrent use of other psychotropic medications at least two weeks prior to baseline
* Concurrent use of other anti-inflammatory medications or anti-cytokine medications. If used on an as-needed (PRN) basis, subjects may enter the study, but will be excluded from cytokine analyses
* Concurrent use of beta-blockers less than one month prior to baseline
* Serious medical illness or instability for which hospitalization may be likely within the next year
* Seizure disorders with the exception of a history of febrile seizures if they occurred during childhood
* Sleep apnea or restless leg syndrome
* Concurrent psychotherapy initiated within 3 months of randomization or ongoing psychotherapy of any duration directed specifically toward treatment of PTSD and/or sleep disturbance
* Patients with significant suicidal ideation
* Current legal actions related to trauma or an ongoing relationship with assailant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pollack, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Center for Anxiety and Traumatic Stress Disorders at Rush, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Eszopiclone: Participants receives 3mg of eszopiclone nightly for 12 weeks, followed by a one month follow-up.
- Placebo: Participants receives 3mg of placebo nightly for 12 weeks, followed by a one month follow-up.
Period: Overall Study
Arm/Group | Eszopiclone | Placebo
Started | 13 | 12
Completed | 7 | 9
Not Completed | 6 | 3
Not completed — Physician Decision | 3 | 2
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eszopiclone | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 8 | 7 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptoms of Post-Traumatic Stress Disorder (PTSD) Between Baseline and Week 12
Description: The Clinician-Administered PTSD Scale (CAPS) is a highly detailed measure of the presence and severity of the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-IV) Post-Traumatic Stress Disorder (PTSD) criteria. The severity score was calculated by adding up the frequency score (scale 0 = "none of the time" to 4 = "most or all of the time") and an intensity score (scale 0 = "none" to 4 = "extreme"), which can then be summed for all 17 symptom questions and/or for the three symptom clusters. Scores range from 0 to 136, where greater than or equal to 80 represents extreme PTSD symptomatology.
Time Frame: Between Baseline and Week 12
Population: Of the 25 subjects that were randomized, 9 did not complete the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 7 | 9
units on a scale | -23 (17.61) | -20 (15.22)

2. Secondary Outcome: Total Score on the Pittsburgh Sleep Quality Index With Post-Traumatic Stress Disorder Addendum (PSQI)
Description: This standard daily sleep diary addresses timing of sleep, ability to fall and stay asleep, dreams, nightmares, and factors which can affect sleep (e.g. caffeine). It requires a summary of the subscales: Duration of sleep + Sleep Disturbance + Sleep Latency + Days of dysfunction due to sleepiness + Sleep efficiency + Overall Sleep Quality + Needing medication to sleep. All subscales are measured from 0 to 3 (Minimum Score = 0 better; Maximum Score = 3 worse). The Minimum TOTAL Score is 0 (better) and Maximum TOTAL Score is 21 (worse).
Time Frame: Changes in total score between Baseline and Week 12 (range of 0 to 21 worse)
Population: Of the 25 subjects that were randomized, 9 did not complete the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 7 | 9
units on a scale | -4.13 (2.93) | -3.33 (3.59)

3. Secondary Outcome: Changes in Emotional Bias Memory Encoding Between Baseline and Week 12
Description: Changes in Emotional Bias Memory Encoding by measuring mean hits minus the false alarms at baseline and at week 12. Subjects perform an encoding session on the 1st day utilizing 147 picture slides, thirty six pictures with negative valence, 36 with neutral valence and additional 75 pictures randomly intermixed. Higher false alarms are associated with lower emotional bias memory encoding.
Time Frame: Baseline and week 12
Population: Subjects with pre treatment and post treatment emotional bias encoding assessments
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 5 | 4
units on a scale | 93 (31) | 102 (32)

4. Secondary Outcome: Cytokine Inflammatory Markers
Description: Differences between baseline and week 12 on Interferon-Gamma, Interleukin-βeta, Interleukin-6, Tumor Necrosis Factor-alpha levels between treatment arms (eszopiclone versus placebo).
Time Frame: Week 12
Population: Subjects with baseline and week 12 cytokine assessments
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Eszopiclone: The total study duration is 16 weeks, with subjects taking 3mg eszopiclone at bedtime for 12 weeks. Cytokine levels were taken at baseline and week 12.
  Eszopiclone: Eszopiclone has been approved by the US Food and Drug Administration (FDA) for the treatment of insomnia (inability to sleep). Eszopiclone has not been specifically approved by the FDA for people who have PTSD-related sleep disturbance.
- Placebo: The total study duration is 16 weeks, with subjects taking placebo at bedtime for 12 weeks. Cytokine levels were taken at baseline and week 12
  Placebo: The placebo used in this study looks exactly like eszopiclone but contains no active ingredients.
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 11 | 10
pg/ml
  Interferon-GAMMA pg/mL | 3.62 (13.98) | -1.55 (6.35)
  Interleukin-βeta pg/mL | -0.10 (4) | 0.30 (7)
  Interleukin-6 pg/mL | 1.29 (8) | -0.08 (9)
  Tumor Necrosis Factor-alpha pg/mL | 67.27 (11) | 64.80 (10)

5. Secondary Outcome: Cytokine Inflammatory Marker on Interleukin-2
Description: Differences between baseline and week 12 on Interleukin-2 levels between treatment arms (eszopiclone versus placebo).
Time Frame: Week 12
Population: Subjects with baseline and week 12 cytokine assessment of Interleukin-2 IU
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 10 | 11
IU | 1.67 (8) | -0.07 (9)

ADVERSE EVENTS:
Arm/Group | Eszopiclone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 9/13 | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eszopiclone (N=13) | Placebo (N=12)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2)
Appetite Increase (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (General disorders) | 1 (1) | 2 (9)
Dysgeusia (General disorders) | 4 (20) | 3 (7)
GI distress (Gastrointestinal disorders) | 2 (5) | 1 (3)
Dizziness (General disorders) | 0 (0) | 1 (2)
Headache (General disorders) | 2 (4) | 3 (5)
Jitteriness (General disorders) | 0 (0) | 1 (2)
Muscle cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Memory impairment (General disorders) | 1 (1) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Urinary hesitation (Renal and urinary disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sedation (General disorders) | 3 (3) | 0 (0)
Sweating (General disorders) | 1 (1) | 0 (0)
Disturbing dreams (General disorders) | 1 (4) | 1 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes